CLINICAL TRIAL: NCT00720759
Title: Improving Stroke Rehabilitation: Spacing Effect and D-cycloserine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B6346-R
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Results first posted 2014-03-07 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-01

CONDITIONS: Stroke
Keywords: stroke; hemiparesis; randomized controlled trial; d-cycloserine; distributed practice; constraint induced movement therapy
MeSH Terms: conditions — Stroke; Paresis | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Experimental): D-cycloserine + distributed treatment
  Interventions: Drug: D-cycloserine + distributed treatment
- Arm 2 (Sham Comparator): D-cycloserine + condensed treatment
  Interventions: Behavioral: D-cycloserine + condensed treatment
- Arm 3 (Placebo Comparator): Placebo + distributed treatment
  Interventions: Drug: Placebo + distributed treatment
- Arm 4 (Placebo Comparator): Placebo + condensed treatment
  Interventions: Behavioral: Placebo + condensed treatment

INTERVENTIONS:
Drug: D-cycloserine + distributed treatment — Subjects will receive CIMT 2 hours/day, 3 days a week, for 10 weeks, in conjunction with d-cycloserine 50 mg PO administered before each treatment session
  Other Names: spaced training
  Arms: Arm 1
Behavioral: D-cycloserine + condensed treatment — Subjects will receive CIMT 6 hours/day, 5 days a week, for 2 weeks, in conjunction with d-cycloserine 50 mg PO administered before each treatment session
  Arms: Arm 2
Drug: Placebo + distributed treatment — Subjects will receive CIMT 2 hours/day, 3 days a week, for 10 weeks, in conjunction with placebo administered before each treatment session
  Other Names: spaced training
  Arms: Arm 3
Behavioral: Placebo + condensed treatment — Subjects will receive CIMT 6 hours/day, 5 days a week, for 2 weeks, in conjunction with placebo administered before each treatment session
  Arms: Arm 4

SUMMARY:
Each year 730,000 Americans experience a stroke. Forty percent are left with significant paralysis of one arm. Certain types of physical therapy, for example constraint induced movement therapy (CIMT), have been shown to be effective in improving arm function. However, for most subjects, improvement is modest. In this trial, we test two approaches that may increase the amount of improvement achieved: 1) distributing treatment over a greater amount of time; and 2) adding a drug, d-cycloserine, which theoretically enhances the molecular mechanisms of learning.

DETAILED DESCRIPTION:
Each year, 730,000 Americans experience a stroke. Forty percent are left with persistent impairment of upper extremity function. Although scientifically vetted rehabilitation therapies for this impairment are starting to emerge, current treatment is generally unsatisfactory. Therapies that seek to engage neuroplastic mechanisms constitute one approach to this problem. A good example is constraint induced movement therapy (CIMT), a treatment that seeks, through extensive functional task practice, to overcome an acquired intentional predisposition to use the spared arm (learned non-use), and to improve motor function in the affected arm. CIMT has been tested in a host of trials, most recently a multicenter randomized controlled trial (RCT) - the EXCITE trial. These trials have generally demonstrated that on average, the treatment shows efficacy, and the results from the RCT indicate that it is more efficacious than "standard" therapies. However, problems with CIMT can be readily identified that pose research challenges: 1) on average, efficacy is limited; 2) only a fraction of subjects show substantial benefit. We propose to address these two problems in a pilot RCT of 20 subjects that will test two modifications of standard CIMT: 1) addition of a drug, d-cycloserine, that may enhance neuroplasticity by potentiating NMDA-glutamate receptor-mediated learning mechanisms; 2) delivery of a fixed amount of CIMT over a greater number of days, which according to learning research, may enhance long-term retention of gains.

All subjects in this trial will receive CIMT. Subjects will be randomized to one of 4 groups:

A. CIMT + d-cycloserine, more condensed treatment B. CIMT + d-cycloserine, less condensed treatment C. CIMT + placebo, more condensed treatment D. CIMT + placebo, less condensed treatment The primary outcome measure will be performance on the Wolf Motor Function Test (time) 3 months after completion of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-80,
* of either sex,
* diverse ethnic background,
* s/p a single unilateral hemispheric stroke 6 or more months prior,
* who meet upper extremity functional criteria for participation in constraint induced movement therapy.

Exclusion Criteria:

* History of more than minor head trauma,
* subarachnoid hemorrhage,
* dementia or other neurodegenerative disease,
* multiple sclerosis,
* lobar intracerebral hemorrhage,
* epilepsy,
* drug or alcohol abuse,
* serious medical illness,
* serum creatinine >1.5,
* schizophrenia,
* major refractory depression,
* insufficient cardiopulmonary function to participate in low-intensity,
* sustained upper extremity exercise,
* severe visual impairment,
* pregnancy,
* inability to understand the potential risks and benefits of the study,
* personally provide informed consent, and
* understand and cooperate with treatment.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen E Nadeau, MD BS BS, Principal Investigator — North Florida/South Georgia Veterans Health System, Gainesville, FL
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited between 1/5/10 and 6/3/11. Recruitment sites included: 1) The VA Rehabilitation Research and Development Brain Rehabilitation Research Center of Excellence at the Malcom Randall VA Medical Center, Gainesville, Florida; and outpatient clinics of the Brooks Rehabilitation Hospital, Jacksonville, Florida.
Pre-assignment Details: All potential participants who met inclusion and exclusion criteria for the study and who provided informed consent were promptly randomized and entered into the study.
Groups:
- Arm 1: D-cycloserine + distributed treatment
  D-cycloserine + distributed treatment : Subjects will receive CIMT 2 hours/day, 3 days a week, for 10 weeks, in conjunction with d-cycloserine 50 mg PO administered before each treatment session
- Arm 2: D-cycloserine + condensed treatment
  D-cycloserine + condensed treatment : Subjects will receive CIMT 6 hours/day, 5 days a week, for 2 weeks, in conjunction with d-cycloserine 50 mg PO administered before each treatment session
- Arm 3: Placebo + distributed treatment
  Placebo + distributed treatment : Subjects will receive CIMT 2 hours/day, 3 days a week, for 10 weeks, in conjunction with placebo administered before each treatment session
- Arm 4: Placebo + condensed treatment
  Placebo + condensed treatment : Subjects will receive CIMT 6 hours/day, 5 days a week, for 2 weeks, in conjunction with placebo administered before each treatment session
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Started | 6 | 6 | 6 | 6
Completed | 6 | 5 | 5 | 6
Not Completed | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 6 | 4 | 4 | 18
  >=65 years | 2 | 0 | 2 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.33 (6.71) | 57.83 (4.40) | 56.50 (12.31) | 58.17 (11.63) | 58.2 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 3 | 2 | 12
  Male | 3 | 2 | 3 | 4 | 12
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 6 | 24

OUTCOME MEASURES:

1. Primary Outcome: Wolf Motor Function Test (Time)
Description: The Wolf Motor Function Test (time) score is the average time in seconds taken to perform each of 15 functional tasks ranging in difficulty from putting one's forearm on a table to stacking checkers. Participants are given 120 seconds to perform a task and if they fail, they are scored 120 for that task. Score range on the WMFT-T is 0-120, lower scores being better.
Time Frame: 3 months after completion of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 6 | 6 | 6 | 6
units on a scale | 10.21 (14.26) | 29.69 (39.06) | 19.09 (32.55) | 26.05 (31.03)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2 vs Arm 3 vs Arm 4; A general linear model was employed. The independent variables were baseline WMFT score, treatment (condensed vs distributed), treatment (d-cycloserine vs placebo), and treatment interaction effect. The dependent measure was WMFT score at 3 months post treatment; Test type: Superiority or Other; p < 0.05, Regression, Linear; Slope = .83, Standard Error of Mean 8.54

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from trial entry through 3 months following treatment completion.
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 1/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 1/6 | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=6) | Arm 2 (N=6) | Arm 3 (N=6) | Arm 4 (N=6)
Recurrent stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=6) | Arm 2 (N=6) | Arm 3 (N=6) | Arm 4 (N=6)
insomnia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
skin tear (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes